CLINICAL TRIAL: NCT03032952
Title: The Efficacy of a Mobile Application for Treating Depression and Anxiety Symptoms in University Students
Brief Title: The Efficacy of a Mobile Application for Treating Depression and Anxiety Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: University of Roehampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8227/001
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Stress, Psychological; Depression; Anxiety
Keywords: RCT; Computerised interventions; Mobile applications; Stress, Psychological; Depressive symptoms; Anxious symptoms; Students; Mental health
MeSH Terms: conditions — Stress, Psychological; Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- "Feel Stress Free" (Experimental): Access to the "Feel Stress Free" mobile application intervention for 12 weeks. Instructed to use it at least once per week for 15 minutes, for the first 6 weeks, then given free access thereafter.
  Interventions: Other: "Feel Stress Free" mobile application
- Wait list control (No Intervention): Given access to the intervention at the end of the 12 weeks of the trial.

INTERVENTIONS:
Other: "Feel Stress Free" mobile application — This online and mobile application uses relaxation techniques, thought challenging, mini-games and mood tracking to help reduce feelings of stress, anxiety and depression.
  Arms: "Feel Stress Free"

SUMMARY:
This was a 12-week, parallel randomised controlled trial, including a 6-week follow-up. The trial compared a group of university students (N = 84) receiving a mobile CBT application intervention ("Feel Stress Free") to a wait-list control group (N = 84) receiving no intervention. Participants were asked to complete the Hospital Anxiety and Depression Scale (HADS) and the Patient Health Questionnaire (PHQ-9) at baseline (as part of the screening questionnaire) and then fortnightly for the 12 weeks. Although blinding was not possible owing to the nature of a wait list control group, researchers did not have any face-to-face contact with the participants, as recruitment and participation in the study was entirely completed online.

DETAILED DESCRIPTION:
This project aimed to test the effectiveness of an application-based computerised Cognitive Behavioural Therapy (cCBT) intervention named "Feel Stress Free" at reducing depression and anxiety symptoms in a sample of UK university students.

This was a 12-week, parallel randomised controlled trial, comparing a group of university students (N = 84) receiving the mobile intervention to a wait-list control group (N = 84) receiving no intervention.

Recruitment took place within the four universities partnered with Thrive UK, all located in London and the South East of England: University College London, University of Roehampton, University of Buckingham and School of Oriental and African Studies (University of London). Recruitment was via the student union or student welfare services of each university, using email advertisements, poster advertisements, personal referrals from student welfare staff, and social media (Twitter and Facebook). The study was conducted entirely online, with all communication between trial personnel and participants via standardised emails.

Participants were instructed to sign up to the trial by navigating to a web page and inserting their email address. They were then sent links to the participant information sheet and consent form. Once they had given their consent, they were sent the screening questionnaire. Randomisation occurred in blocks of 30 - each time 30 eligible participants had completed the screening questionnaire, they were randomised by an independent statistician, with an equal number of participants allocated to each arm.

Participants in the intervention group received a link to download the "Feel Stress Free" application free of charge, and participants in the control group were informed that they would receive access to the application when the trial was over. Those in the intervention group were asked to use the app at least once per week for 15 minutes for the 6 weeks of the main trial, and then as often as preferred for the follow-up period. The "Feel Stress Free" application consists of relaxation activities such as breathing exercises, progressive muscle relaxation and meditation, as well as relaxing mini-games, uplifting messages and negative thought tracking. Users are prompted daily to measure and track their mood, and activity recommendations are given if needed.

All participants were asked to complete the Hospital Anxiety and Depression Scale and Patient Health Questionnaire fortnightly for the 12 weeks, with the screening questionnaire taken as 'week 0'. They were sent reminders throughout the week if they did not do so. The HADS is a measure of the severity of anxiety and depression symptoms that an individual is experiencing, and the PHQ is a measure of the severity of depression symptoms an individual is experiencing. Both are suitable for use in the general population.

All questionnaires were completed via a secure email link, using Participant IDs assigned at the beginning of the trial. All data were anonymised when stored, and each participant was provided with a contact email address, which was used to seek help regarding the study or to withdraw. Whilst it was not possible to blind trial personnel, owing to the nature of a wait list control group, there was no face-to-face or personalised contact between trial personnel and participants, unless a participant sent a query email.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Provided informed consent
* Self-identified as often feeling anxious or depressed, and scored 8 or above on one or both subscales of the HADS (indicating at least possible caseness)
* Currently a student at one of the four partnered universities
* Had access to an Apple or Android phone or tablet, or a computer with Firefox, Safari or Chrome installed
* Able to use the aforementioned device (computer literacy)

Exclusion Criteria:

* Failure to provide a valid email address for one of the four partnered universities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2016-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | At baseline and then fortnightly for 12 weeks
  A self-report measure comprised of 2 subscales, one for depression and one for anxiety.

SECONDARY OUTCOMES:
1 Patient Health Questionnaire (PHQ-9) | At baseline and then fortnightly for 12 weeks
  Self-report measure of depression used in UK primary care

CONTACTS AND LOCATIONS:
Overall Officials: Andres Fonseca, MBBS, MSc, Principal Investigator — University College, London; Tayla L McCloud, MSc, Study Director — University College, London; Elias Tsakanikos, PhD, Principal Investigator — University of Roehampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCloud T, Jones R, Lewis G, Bell V, Tsakanikos E. Effectiveness of a Mobile App Intervention for Anxiety and Depression Symptoms in University Students: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Jul 31;8(7):e15418. doi: 10.2196/15418. PMID 32735221